CLINICAL TRIAL: NCT02288546
Title: Vegans Exposure to Pesticides and Nitrate
Brief Title: Vegans Health Status and Exposure to Pesticides and Nitrate
Status: Completed | Type: Observational
Sponsor: University of Eastern Finland (Other)
Collaborators: Finnish Institute for Health and Welfare (Other Government); Helsinki University Central Hospital (Other); Finnish Safety and Chemicals Agency (Unknown)
Responsible Party: Sponsor
Other Study IDs: UKuopio
Record Dates: First submitted 2014-11-03; First posted 2014-11-11 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2011-08

CONDITIONS: Malnutrition
Keywords: nutritional status; pesticides; nitrate
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vegans: Vegans' data are compared with those of sex-and age-matched non vegetarians
- Non-vegans: Non-vegans are age and sex-matched controls

SUMMARY:
This research concerns nutritional and toxicological health risk evaluation among long-term vegans. Research focus is in cumulative exposure to pesticides.

DETAILED DESCRIPTION:
The main objective of the study was nutritional and toxicological health risk evaluation among long-term vegans with emphasis on cumulative exposure to pesticides. Main research methods include: measurement of food intake by using three days food record, measurement of nutritional and toxicological bio-markers on blood, serum and plasma. Nutritional biomarkers include following plasma/ serum measurements: concentrations of vitamins (vitamin E, D2, D3, B12 and beta-carotene), iron, iodine, selenium, fatty acids and polyphenols. Toxicological measurements include nitrate, pesticides and DNA-adducts.

We recruited the participants (n = 41) through an advertisement published in the Finnish Vegan Association's monthly newspaper and via an online discussion forum. The selection criteria were as follows: the participants had to (1) have followed a vegan diet for at least a year, (2) be between 18 and 50 years of age, (3) be apparently healthy, and (4) be nonusers of regular medications (except oral contraceptives or hormone replacement therapy). Further, we matched the non-vegetarian participants by age and sex. The study was approved by the Ethical Committee of Kuopio University Hospital (69//2011)

We assessed the consumption of foods at baseline with a three-day food record using household measures. The participants received the instructions on how to complete this record, and a dietician checked the completed food records. The participants also filled out a health questionnaire inquiring into their long-term healthy eating habits, including vitamin supplementation.

We collected fasting peripheral venous blood samples, plasma and serum, and stored them at -70 °C before the analysis. Further, urine samples 24 hours were collected prior to phlebotomy and divided into aliquots. For one of the subjects, only a spot urine sample was available. We carried out the hematological and chemical analyses at laboratory (hematological data), Helsinki University Central Hospital (folate, vitamin B12, vitamin D, and homocysteine), and the National Institute for Health and Welfare (alfa-tocopherol, beta-carotene, selenium, iodine, fatty acid profile, and polyphenols). Nitrate, nitrite were measured by capillary electrophoresis and DNA adducts by ELISA at Finnish Food Safety Authority.

ELIGIBILITY:
Inclusion Criteria:

The selection criteria were as follows: the participants had to

1. have followed a vegan diet for at least a year,
2. be between 18 and 50 years of age,
3. be apparently healthy, and
4. be nonusers of regular medications (except oral contraceptives or hormone replacement therapy). Further, we matched the non-vegetarian participants by age and sex.

Exclusion Criteria:

* age <18, and >50y,
* regular medication,
* illnesses

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Vegans and non-vegans
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Nutritional and toxicological status (determined by measuring several nutritional biomarkers from blood and urine) | 1 year
  Nutritional status was determined by measuring several nutritional biomarkers (vitamin E, D2,D3, B12, , beta-carotene, iron, iodine, selenium, fatty acids, polyphenols) from serum/plasma or urine

SECONDARY OUTCOMES:
Food intake (recorded by 3-day records) | 3 days
  Food intake was recorded by 3-day records
Nitrate excretion (urinary nitrate determination) | 24 hr
  urinary nitrate determination

CONTACTS AND LOCATIONS:
Overall Officials: Anna-Liisa Kosonen, PhD, Principal Investigator — University of Eastern Finland
Locations (1):
- University of Eastern Finland, Kuopio, Finland, Finland